CLINICAL TRIAL: NCT03910933
Title: EKITE: Electronic KIDCLOT Interactive Thrombosis/Thrombophilia Education; A Quality Assurance Initiative
Brief Title: Electronic KIDCLOT Interactive Thrombosis/Thrombophilia Education; A Quality Assurance Initiative
Acronym: eKITE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00074672
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Health Literacy; Anticoagulation
Keywords: Warfarin; Child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: elearning patient information — The videos will standardize patient teaching about anticoagulants, warfarin, INR testing, and warfarin safety for Patient Self-Testing, and Patient Self-Management. eKITE, will provide a user-friendly interface to provide health education about anticoagulation. eKITE will teach concepts to the patient, facilitate sustained patient knowledge (6 month evaluation), reduce stress associated with learning, actively engage patients in their anticoagulant management (preference, satisfaction and knowledge).

SUMMARY:
Effective patient education improves health literacy and engagement thus improving long-term health outcomes. Health literacy is imperative to make informed health decisions and relies on the ability to obtain, process and understand health information; and is the cornerstone of safe health management. It is necessary to evaluate educational initiatives to determine their effectiveness in knowledge translation.

A more effective way to provide patient education is to utilize media technology. Current education styles do not teach patients in the best way as they are not consistent with how people of all ages currently learn (through technology). In addition, patient teaching most commonly occurs during highly stressful times like hospital visits with new diagnoses. Current patient educational methods are costly given the amount of health provider time required.

Electronic KITE teaching modules are infographic visual representations that present information quickly and clearly, integrating words and graphics to tell a story to reveal information. Infographic presentations are tools which facilitate self-directed learning with understandable, accessible information presented in an engaging way with an aim to enhance learning for children and their families. Patients are able to learn at a pace consistent with their learning style to facilitate knowledge development and health literacy.

DETAILED DESCRIPTION:
A more effective way to provide patient education is to utilize media technology. Current education styles do not teach patients in the best way as they are not consistent with how people of all ages currently learn (through technology). In addition, patienteaching most commonly occurs during highly stressful times like hospital visits with new diagnoses. Current patient educational methods are costly given the amount of health provider time required.

Electronic KITE teaching modules are infographic visual representations that have been developed to provide patient teaching related to warfarin and its management.

How much patients have learned will be assessed using the KIDCLOT validated knowledge quizzes. Children 8 years and older to have cognitive capacity will complete the quizzes if able. Caregivers will complete all quizzes linked with the modules they have completed.

Patients may be enrolled into the appropriate cohort based on the health provider decision for management.

1. Warfarin international normalized ratio (INR) testing
2. Warfarin with home INR testing
3. Warfarin transition from home INR testing to warfarin self management.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients and their caregivers who are receiving treatment with anticoagulant therapy.

Exclusion Criteria:

* Non-english speaking patients.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: English speaking children and their caregivers who initiate or require ongoing anticoaogulant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
KIDCLOT What is an Anticoagulant Quiz1 | enrolment
  Quiz to assess patient learning of important concepts related to anticoagulants
KIDCLOT What is an Anticoagulant Quiz1 | 6 months and 18 months
  Quiz to assess change in patient knowledge of important concepts related to anticoagulants
Kidclot Warfarin Quiz 2 | enrolment
  Quiz to assess patient learning of important concepts related to warfarin
Kidclot Warfarin Quiz 2 | 6 months and 18 months
  Quiz to assess patient learning of important concepts related to warfarin
KIdclot INR testing Quiz 3 | enrolment
  Quiz to assess patient learning of important concepts related to INR testing
KIdclot INR testing Quiz 3 | 6 and 18 months
  Quiz to assess change in patient knowledge of important concepts related to INR testing
Kidclot safety on an anticoagulant Quiz 4 | enrolment
  Quiz to assess patient learning of important concepts related to patient safety on an anticoagulant
Kidclot safety on an anticoagulant Quiz 4 | 6 months and 18 months
  Quiz to assess change in patient knowledge of important concepts related to patient safety on an anticoagulant
Kidclot Home INR testing Quiz 5 | enrolment
  Quiz to assess patient learning of important concepts related to home INR testing
Kidclot Home INR testing Quiz 5 | 6 and 18 months
  Quiz to assess change in patient knowledge of of important concepts related to home INR testing
Kidclot Warfarin Self Management Quiz 6 | 6 months
  Quiz to assess patient learning of important concepts related to Warfarin Self Management
Kidclot Warfarin Self Management Quiz 6 | 18 months
  Quiz to assess change in patient knowledge of of important concepts related to Warfarin Self Management

SECONDARY OUTCOMES:
Patient preference | enrolment
  Questionnaire
Stress Around Learning Score STAI-1 | enrolment
  Survey to Assess patient stress around learning about warfarin and its management using the on-line modules. Measure of Calm.- Total score out of 40 with higher score indicates low stress and a positive outcome
Stress Around Learning Score STAI-1 | enrolment
  Survey to Assess patient stress around learning about warfarin and its management using the on-line modules. Total score out of 40. Measure of Worry- Total score out of 40 with lower score indicates low stress indicating a positive outcome
Pediatric Anticoagulation Quality of Life | 6
  Quality of life score to assess impact of warfarin therapy on health related quality of life. Lower score indicates low impact. Score is a percentage
Pediatric Anticoagulation Quality of Life | 18 months
  Quality of life score to assess any change in impact of warfarin therapy on health related quality of life. Lower score indicates low impact. Score is a percentage

OTHER OUTCOMES:
Time in therapeutic Range | 18 months
  Time INRs are within range
Health care provider time associated with warfarin teaching | enrolment, 6 months and 18 months
  Providers will measure and report the additional time spent providing patient teaching for warfarin management

CONTACTS AND LOCATIONS:
Overall Officials: Mary Bauman, MN, Principal Investigator — Stollery Children's Hospital, University of Alberta
Locations (6):
- United States (4):
  - Ann & Robert H Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Texas Children'Hospital, Houston, Texas
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital of Easter Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No